CLINICAL TRIAL: NCT02169232
Title: Videolaryngoscope Versus Fiberoptic Bronchoscope for the Awake Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Albert Moore, Assistant professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13-443-SDR
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Need of Awake Intubation for Difficult Airways
Keywords: Awake intubation; Videolaryngoscope; Fiberoptic
MeSH Terms: interventions — Optical Fibers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Videolaryngoscope (Active Comparator): Intubation by videolaryngoscope
  Interventions: Device: Videolaryngoscope
- Fiberoptic (Active Comparator): Intubation by fibroscope
  Interventions: Device: Fiberoptic

INTERVENTIONS:
Device: Videolaryngoscope
  Other Names: Intubation by Glidoscope
  Arms: Videolaryngoscope
Device: Fiberoptic
  Arms: Fiberoptic

SUMMARY:
Endotracheal intubation of the morbidly obese is often performed awake. Fiberoptic bronchoscope assisted endotracheal intubation, a commonly utilized technique for securing an airway while a patient is awake, has many limitations. The video laryngoscope is a device that is similar to a conventional laryngoscope but uses a video system to visualize the larynx. Because of its low cost, ease of use, and usefulness in the presence of edema or bleeding that may obstruct the airway, video assisted laryngoscopy has been shown to be useful for awake endotracheal intubations. However, a direct comparison of the fiberoptic bronchoscope with video assisted laryngoscopy has not been performed for awake endotracheal intubations in of obese patients. Patients undergoing laparoscopic gastric bypas andrecquiring awake intubations will be randomized for either fiberoptic bronchoscope or video assisted laryngoscopy. The investigators primary outcome will be the time required for successful intubation.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patient presenting for bariatric surgery at the Royal Victoria Hospital

Exclusion Criteria:

* moderate to severe systemic illness, i.e. American Society of Anesthesiologists (ASA) score of 4 or higher
* inability to communicate in English or French
* contraindications to the drugs used in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The time required for successful intubation | 10 minutes
  The time required for successful intubation, which will be measured as the time from which the bronchoscope or videolaryngoscope is initially introduced into the oropharynx, until the time that CO2 is registered on the capnogram.

SECONDARY OUTCOMES:
Number of intubation attempts, defined as a complete withdrawal and re-insertion of the airway instrument. | 10 minutes

OTHER OUTCOMES:
The ease of intubation using a 10 cm visual analogue scale, completed both by the person performing the intubation, and an independent observer. | one hour
Post-operatively the patient's satisfaction | 24 hours
  Post-operatively the patient's satisfaction with the procedure using a 10 cm visual analogue scale, a discomfort scale using a 10 cm visual analogue scale, whether they would recommend this procedure to a future patient, and the severity of sore throat using a 10 cm visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Moore, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada